CLINICAL TRIAL: NCT06376786
Title: Italian iTTP Registry (a Prospective Observational Study)
Brief Title: Italian iTTP Registry
Status: Recruiting | Type: Observational
Sponsor: Fondazione Luigi Villa (Other)
Responsible Party: Sponsor
Other Study IDs: ItaliTTP
Record Dates: First submitted 2024-03-15; First posted 2024-04-19 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-04

CONDITIONS: TTP - Thrombotic Thrombocytopenic Purpura
Keywords: ADAMTS13; Thrombotic microangiopathy
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic; Thrombotic Microangiopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- iTTP patients: iTTP patients will be treated and followed-up as per standard clinical practice.

SUMMARY:
ItaliTTP is an observational, prospective, single-arm, national, multicenter, non-pharmacological cohort study aimed at better defining and understanding the natural history, disease severity, and clinical outcomes of patients with immune-mediated thrombotic thrombocytopenic purpura (iTTP) in Italy.

A minimum of 132 consecutive patients with acute iTTP (first event or relapse) will be enrolled for 3 years, with the possibility of extension, with a follow-up period of 3 years.

DETAILED DESCRIPTION:
Acquired immune-mediated thrombotic thrombocytopenic purpura (iTTP) is a rare, life-threatening thrombotic microangiopathy characterized by episodes of thrombocytopenia, microangiopathic hemolytic anemia, and extensive microvascular thrombosis leading to multiorgan involvement. Despite advances in understanding iTTP etiology and management in the acute phase, significant gaps in knowledge about its progression, particularly during clinical remission and concerning long-term complications, persist.

ItaliTTP, a national, multicenter, observational, prospective, non-pharmacological cohort study, aims to elucidate the natural history, severity, and outcomes of iTTP in Italy. The study will enroll hospitalized iTTP patients (experiencing either initial or recurrent episodes) and follow them in outpatient settings across participating Italian centers. The study plans to include at least 132 patients of any gender, aged 12 to 99, over a three-year period, with an option for extension, and a three-year follow-up. During hospitalization and subsequent outpatient visits, participants will undergo routine clinical assessments and laboratory tests. In addition to these data, peripheral blood samples will be collected for ADAMTS13 analysis and potential future research.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an acute iTTP episode (first event or relapse), defined by thrombocytopenia and microangiopathic hemolytic anemia, in the absence of alternative causes, and the presence of severe deficiency of ADAMTS13 activity (< 10 IU/dL or <10% of normal value) and anti-ADAMTS13 autoantibodies
* Both male and female patients, aged 12 years or older
* Patients who have signed the informed consent for the participation to the study

Exclusion Criteria:

* Patients who have not signed the informed consent for the participation to the study

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients with an acute event of iTTP (first event or relapse), then followed-up in outpatient clinics of the participating centers.
Sampling Method: Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Age at onset | 3 years
  Age at the first acute iTTP episode in years
Sex | 3 years
Birth Country/Region | 3 years
Race | 3 years
Blood group | 3 years
  ABO/Rh blood group
BMI | 3 years
  Body mass index in kg/m^2
Proportion of patients with comorbidities, including: autoimmune diseases, cancer, HIV infection, hypertension, type 2 diabetes, hypercholesterolemia, cardiovascular disease, chronic renal failure, liver disease, depression. | 3 years
  Proportion of iTTP patients with comorbidities
Proportion of acute iTTP episodes preceded by potential triggering factors including: infections, pregnancy, surgery, psychological trauma, vaccination, drugs | 3 years
  Proportion of potential triggering conditions/events/drugs occured/taken in the 3 months prior the acute iTTP episode
Incidence, type and severity of clinical manifestations, including: bleeding, cardiovascular, neurological, renal and systemic signs and symptoms | 3 years
  Incidence, type and severity of clinical manifestations at presentation of the acute iTTP episode
Platelet count lactate dehydrogenase (LDH), total and indirect bilirubin, liver transaminases, creatinine, troponin | 3 years
  Platelet count at presentation of the acute iTTP episode, expressed in number x 10^9/L
Hemoglobin lactate dehydrogenase (LDH), total and indirect bilirubin, liver transaminases, creatinine, troponin | 3 years
  Hemoglobin level at presentation of the acute iTTP episode, expressed in g/dL
Lactate dehydrogenase (LDH) lactate dehydrogenase (LDH), total and indirect bilirubin, liver transaminases, creatinine, troponin | 3 years
  LDH level at presentation of the acute iTTP episode, expressed in IU/L
Creatinine lactate dehydrogenase (LDH), total and indirect bilirubin, liver transaminases, creatinine, troponin | 3 years
  Creatinine level at presentation of the acute iTTP episode, expressed in mg/dL
Cardiac troponin | 3 years
  Cardiac troponin level at presentation of the acute iTTP episode, expressed in ng/L
ADAMTS13 activity | 6 years
  Level of functional ADAMTS13 activity expressed in IU/dL or %
Anti-ADAMTS13 antibodies | 6 years
  Concentration or presence/absence of anti-ADAMTS13 antibodies
Number of daily therapeutic plasma exchange procedures | 3 years
  Number of daily therapeutic plasma exchange procedures to achieve clinical response of the acute iTTP episode
Proportion of acute iTTP patients treated with rituximab | 6 years
Proportion of acute iTTP patients treated with immunosuppressors other than steroids and rituximab | 6 years
Proportion of iTTP patients treated with caplacizumab | 3 years
Incidence, type and severity of TTP-related drugs adverse events | 6 years
  Incidence, type and severity of TTP-related drugs adverse events recorded during the acute iTTP episode and disease remission of iTTP patients
Proportion of iTTP patients achieving clinical remission | 6 years
  Proportion of iTTP patients achieving clinical remission defined as sustained clinical response with either no therapeutic plasma exchange (TPE) and no anti-von Willebrand factor (VWF) therapy for ≥ 30 days or with attainment of ADAMTS13 remission, whichever occurs first.
Proportion of iTTP patients refractory to acute iTTP treatment | 6 years
  Proportion of iTTP patients refractory to acute iTTP treatment. Refractoriness defined as persistent thrombocytopenia and a persistently raised LDH level despite treatment.
Proportion of iTTP patients experiencing complications during hospitalization, including: bleeding, thrombosis, neurological, renal, cardiac complications | 6 years
  Proportion of patients who experience complications during the hospitalization for acute iTTP
Proportion of iTTP patients experiencing clinical exacerbation | 6 years
  Proportion of iTTP patients experiencing clinical exacerbation defined as sustained platelet count ≥ 150 × 109/L (or above the local lower limit of normal [LLN]) and LDH < 1.5 times hte upper limit of normal (ULN) and no clinical evidence of new or progressive ischemic organ injury.
Proportion of iTTP patients achieving ADAMTS13 remission | 6 years
  Proportion of iTTP patients achieving ADAMTS13 remission defined as ADAMTS13 activity ≥ 20% to < LLN (partial) or ADAMTS13 activity ≥ LLN (complete).
Time to clinical response | 6 years
Time to clinical remission | 6 years
Time to ADAMTS13 remission | 6 years
Proportion of iTTP patients with a clinical relapse | 6 years
  Proportion of iTTP patients with a clinical relapse defined as a platelet count decrease to < 150 × 109/L (with other causes of thrombocytopenia ruled out), with or without clinical evidence of new ischemic organ injury, after a clinical remission.
Proportion of iTTP patients with an ADAMTS13 relapse | 6 years
  Proportion of iTTP patients with an ADAMTS13 relapse defined as a decrease of ADAMTS13 activity to < 20% after a partial or complete ADAMTS13 remission.
Time to clinical relapse | 6 years
Time to ADAMTS13 relapse | 6 years
Incidence, type and severity of pregnancy complications in iTTP pregnant women | 6 years

SECONDARY OUTCOMES:
iTTP incidence in Italy | 3 years
  The number of all TTP events (first events and relapses) and first TTP events will be divided by the number of people at risk multiplied by the observation time to estimate the incidence rate of iTTP events and iTTP incident cases, respectively (in persons-years).

CONTACTS AND LOCATIONS:
Overall Officials: Flora Peyvandi, MD, PhD, Principal Investigator — Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milano, Italy
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, MI, Italy